CLINICAL TRIAL: NCT06528626
Title: Wedge-Shaped Clusterded Randomizad Trial to Evaluate Two Tools to Identify People At Risk or Already Infected with HIV and HCV
Brief Title: Tools to Identify People At Risk or Already Infected with HIV and HCV
Acronym: ATENEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: PI22/01878
Record Dates: First submitted 2023-07-05; First posted 2024-07-30 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-07

CONDITIONS: HIV/AIDS; STD; HCV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Observational (No Intervention)
- self-questionnaire SQ-R&IC (Active Comparator)
  Interventions: Diagnostic Test: rapid HIV and HCV serological tests
- rapid HIV and HCV serological tests (Active Comparator)
  Interventions: Diagnostic Test: rapid HIV and HCV serological tests

INTERVENTIONS:
Diagnostic Test: rapid HIV and HCV serological tests — In the standard of care branch (SOC), the health personnel will ask people a series of questions to identify the HIV risk exposition, and also they will be provided pop-up computer alerts of HIV indicator conditions in the electronic medical record, moreover HIV and HCV serological tests will be carried out in the reference laboratory, while in the intervention branch in addition to the SOC, a SQ-R&IC of HIV and HCV will be made available to the HC population, through a quick response (QR) code, as well as HIV and HCV RT.
  Other Names: self-questionnaire SQ-R&IC
  Arms: rapid HIV and HCV serological tests; self-questionnaire SQ-R&IC

SUMMARY:
Wedge-Shaped Clusterded Randomizad Trial to Evaluate Two Tools to identify People at Risk or already Infected with HIV and HCV

DETAILED DESCRIPTION:
Objectives: To reduce hidden and incident HIV and HCV infection, through the implementation of a risk and indicator conditions self-questionnaire SQ-R&IC for HIV and HCV infection, in addition to rapid HIV and HCV serological tests (RT), in the Health Centers (HC). Methodology: stepped-wedge cluster randomized trial in 8 CS of the community of Madrid, to to know if the implementation of the 2 tools described above, improve risk identification and subsequent screening for HIV and HCV infection. In the standard of care branch (SOC), the health personnel will ask people a series of questions to identify the HIV risk exposition, and also they will be provided pop-up computer alerts of HIV indicator conditions in the electronic medical record, moreover HIV and HCV serological tests will be carried out in the reference laboratory, while in the intervention branch in addition to the SOC, a SQ-R&IC of HIV and HCV will be made available to the HC population, through a quick response (QR) code, as well as HIV and HCV RT. The variables that will be compared are the percentage of HIV and HCV tests performed, of people referred to receive PrEP, and of new HIV and HCV diagnoses or not linked to care that are made during the periods assigned to the EDC branch vs. those in the intervention branch.

ELIGIBILITY:
Inclusion Criteria:

- 14-65 years in the health area or who are captured for inclusion by health personnel. They give their consent to participate.

Exclusion Criteria:

* Having already been included in the study, not signing the consent.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Implementation of a risk and indicator conditions self-questionnaire SQ-R&IC for HIV and HCV infection, in addition to rapid HIV and HCV serological tests | 3 years
  Number of Participants With the implementation of a risk and indicator conditions self-questionnaire SQ-R&IC for HIV and HCV infection, in addition to rapid HIV and HCV serological tests, Change From Baseline in hidden and incident HIV and HCV infection at 3 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Maria J. Vivancos-Gallego, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No